CLINICAL TRIAL: NCT02863640
Title: Evaluation of the Protective Role of the L-DOPA Against Age Related Macular Degeneration in Parkinson's Patients
Acronym: PARM
Status: Terminated | Type: Observational
Why Stopped: Major difficulties of patient inclusions
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2015_33
Record Dates: First submitted 2016-08-03; First posted 2016-08-11 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Macular Degeneration, Senile
Keywords: Senile macular degeneration; Parkinson's disease
MeSH Terms: conditions — Macular Degeneration, Age-Related, 2; Macular Degeneration; Parkinson Disease | interventions — Tomography, Optical Coherence; Optical Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Exposed patients: Patients treated for Parkinson's disease with a cumulative dose of L-DOPA above the 59th percentile of the population
  Interventions: Device: Color retinography; Device: Optical coherence tomography; Device: Fundus autofluorescence imaging
- Non exposed patients: Patients treated for Parkinson's disease with a cumulative dose of L-DOPA below the 41th percentile of the population
  Interventions: Device: Color retinography; Device: Optical coherence tomography; Device: Fundus autofluorescence imaging

INTERVENTIONS:
Device: Color retinography
Device: Optical coherence tomography
Device: Fundus autofluorescence imaging

SUMMARY:
Age related macular degeneration (ARMD) is a major and irreversible cause of blindness among the elderly. The sub-retinal space, located between the retinal pigmentary epithelium (RPE) and the external segments of the retinal photoreceptors, plays a crucial role in this pathology. A recent epidemiologic study in the US, unpublished yet, has shown that patients treated with the L-DOPA, developed only later an ARMD when compared to the untreated patients.

The L-Dopa is an endogenous ligand of the GPR43 receptor, located on the RPE's cell's apical pole.

This receptor, via several intracellular mechanisms, regulates the cell's exosomal and endosomal pathways: it would appear that the L-DOPA, by stimulating this receptor, decreases significantly the RPE's exosome release.

The contents of the exosomes is still uncertain, however in addition to their signalization role, it seems they transport pro-inflammatory components, possibly helping the cellular recruitment due to the mononuclear phagocytic systems, particularly toxic for the photoreceptors.

The aim of this study is to validate the hypothesis stating that he L-DOPA would play a protective role against age related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged of 70 years old and more
* Parkinson's disease

Exclusion Criteria:

* Opposition to participate in this trial
* Patient under a measure of legal protection
* Absence of affiliation to social security or universal health coverage (CMU)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Population of patients followed at Rothschild's Ophthalmologic Foundation for Parkinson's disease.
  The study is proposed to patients aged of 70 years old and more and with a cumulative dose of L-DOPA above the 59 th percentile of the population or with with a cumulative dose of L-DOPA below the 41th percentile of the population
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Diagnosis of ARMD based on ophtalmological examination combining color retinography, optical coherence tomography and fundus autofluorescence Imaging | Diagnosis of ARMD made during a single consultation lasting about an hour
  Risk of ARMD : Ratio between the ARMD prevalence rate in patients with an elevated cumulated dose of L-DOPA and the ARMD prevalence rate in patients with a low cumulated dose of L-DOPA Risk adjusted according to age and sexe

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A. de Rotchschild, Paris, France